CLINICAL TRIAL: NCT00862927
Title: Cue Reactivity in Virtual Reality: The Role of Context
Status: Terminated | Type: Observational
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0544
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Smoking
Keywords: Smoking Cessation; Cigarette Smoking; Tobacco Smoking; Cue Reactivity; Virtual Reality; VR; Contextual Cues; Explicit Smoking Cues; Craving; Physiological Arousal; Nicotine Dependence; Breath Sample; Saliva Test; Questionnaire
MeSH Terms: conditions — Smoking; Smoking Cessation; Cigarette Smoking; Tobacco Smoking; Tobacco Use Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cue reactivity in virtual reality: Breath Scan + Saliva Sample + Questionnaires + View Virtual Reality Scenes
  Interventions: Other: Breath Sample; Other: Saliva Sample; Behavioral: Questionnaire; Behavioral: View Virtual Reality Scenes

INTERVENTIONS:
Other: Breath Sample — Breathe into machine measuring carbon monoxide.
Other: Saliva Sample — Chew cotton ball for 30 seconds for cotinine measurement.
Behavioral: Questionnaire — 6 surveys, taking approximately 30 minutes total.
Behavioral: View Virtual Reality Scenes — Use virtual reality helmet and hand-held controller to answer questions about 4 viewing scenes while wearing physiological measurement skin sensors, approximately 6 minutes.
  Other Names: VR

SUMMARY:
The objectives of this proposal are to examine the role of context in a virtual reality (VR) environment and to explore the extent to which cues (i.e., contextual cues or explicit smoking cues) influence craving and physiological arousal within VR.

The current study seeks to determine whether smokers, placed in the context of a VR convenience store devoid of explicit smoking cues, will experience less craving and physiological arousal, compared to exposure to the same VR environment containing explicit smoking cues. This important line of inquiry will help clarify the influence of environmental contexts that may contribute to the overall reactivity effects (e.g., craving, arousal) smokers experience when confronted with cues associated with smoking.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete a breath scan test, a saliva sample, complete questionnaires, smoke 1 cigarette, have your physiological measurements recorded, and view virtual reality scenes.

Breath Sample:

After signing the consent form, you will be asked to provide a breath scan to show how recently you smoked. To provide a breath sample, you will hold your breath for 15 seconds and exhale (breathe out) through a small cardboard tube into a small machine. This machine measures the amount of carbon monoxide in your breath, which provides an estimate of how many cigarettes you have recently smoked. If this measurement shows you are a very light smoker, you may not be able to take part in the rest of this study.

Saliva Sample:

You will be asked to provide a saliva sample in order to measure cotinine, which is a substance related to nicotine that is found in the body after smoking recently. You will be asked to place a small cotton roll in your mouth and gently chew the roll for 30 seconds. You will then remove the roll and place it in a small container. The container will not be labeled with your name, but only a study ID number. Only the study staff will have access to this number. Once the samples have been measured for levels of cotinine, the samples will be destroyed.

Questionnaires:

You will fill out a questionnaire that includes questions about your age, smoking history, marital status, ethnicity, and other basic information. This questionnaire should take about 3 minutes to complete. You will also complete 5 additional questionnaires that will ask about your mood, thoughts and feelings, and smoking behavior. These questionnaires should take about 30 minutes total to complete.

While completing the questionnaires, you will be asked to smoke 1 cigarette (any brand). You will be told to bring in your own cigarettes for this part of the study. However, if you forget to bring them in, the study staff will be able to provide one to you. This will be done so that all participants will have smoked their last cigarette at about the same time before viewing the virtual reality scenes.

Physiological Measurements:

Your heart rate and the amount you sweat will be recorded after completing the questionnaires and during each virtual reality scene (described below) by applying small sensors to your skin.

After you have completed the questionnaires, you will sit in a recliner and the sensors will be placed on your rib cage and hand. The sensors that measure heart rate will be placed in the following locations: your lower left rib cage, just under your right collar bone, and just under your left collar bone. The sensors that measure the amount you sweat will be placed on the palm of your hand.

The Virtual Reality Scenes:

You will sit in a recliner and be asked to put on a virtual reality helmet, which has goggles and noise-cancelling headphones. You will be told how to wear the helmet and use the hand-held controller to answer the questions you will see after you have finished viewing each virtual reality scene.

You will view 2 virtual reality scenes that will either show images of nature, such as fish, or images of a convenience store, such as a parking lot of a gasoline station and the inside of store. The experience of virtual reality may involve other senses as well. For example, you may hear, smell, and feel sensations (such as mild vibrations) that are associated with the scenes you are viewing.

After each virtual reality scene that you view, you will answer a single question about your desire to smoke. It should take less than 1 minute to complete the question. You will view two virtual reality scenes, with a five minute rest period in between. It will take about 6 minutes to view each pair of scenes. After the scenes have ended, the equipment and sensors will be removed, and you will be asked to complete a questionnaire that will ask about your experiences and feelings about virtual reality. This questionnaire should take less than 10 minutes to complete.

Length of Study:

Once you have finished viewing the virtual reality scenes and completed the last questionnaire, your participation in this study will be over. Your total participation time in this study should take about 90 minutes.

This is an investigational study. Up to 75 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Self-report of smoking at least 10 cigarettes per day
3. Expired carbon monoxide (CO) equal to or greater than 10 ppm
4. English speaking and able to read at > 6th grade level
5. Not interested in quitting smoking in next 30 days

Exclusion Criteria:

1) Self-report history of motion sickness or vertigo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers, 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Differences in craving and arousal among four scenarios based on repeated survey measure | Total participation time about 90 minutes; Overall study period (assessment & surveys) approximately 2 years
  Analyses on craving and arousal measures between-subjects to discern any differences in craving and arousal among the two sets of scenarios. After providing breath and saliva samples, seated participants complete questionnaires and smoke one cigarette to control for variability in time since last cigarette. First 5 questionnaires take approximately 35 minutes to complete, and another, completed after the VR session, approximately 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Brian L. Carter, PhD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org